CLINICAL TRIAL: NCT04761510
Title: Mindfulness-SOS: Stress Reduction for Refugees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mindfulness-SOS for Refugees
Record Dates: First submitted 2021-01-12; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-02

CONDITIONS: Stress Disorders, Post-Traumatic; Stress Related Disorder
Keywords: Forcibly Displaced Persons; Post-migration Stress; Trauma; Post-traumatic Stress Disorder; Depression; Anxiety; COVID-19 Pandemic; Stress; Online Mental Health Intervention Program; Treatment Adherence; Mindfulness; Compassion
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Depression; Anxiety Disorders; COVID-19; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Mindfulness-SOS for Refugees — Mindfulness-SOS for Refugees is a brief internet-based mobile-supported intervention program which is a mobile-health adaptation of MBTR-R - a mindfulness- and compassion-based, trauma-sensitive, and socio-culturally adapted group intervention program designed for FDPs. Mindfulness-SOS for Refugees entails 8 brief sessions and 9 mindfulness meditation practice exercises - delivered via audio recordings using participants' smartphones. The intervention program is specifically designed to mitigate acute stress and related mental health symptoms among FDPs. During participation in the Mindfulness-SOS for Refugees intervention program, participants will be encouraged to complete 2 sessions per week and practice each day for 4 weeks but can choose to extend this up to 8 weeks. Delivery of Mindfulness-SOS for Refugees entails administrative guidance as well as adherence-focused guidance.

SUMMARY:
The COVID-19 pandemic crisis is associated with a wide range of stressors for the general population. For forcibly displaced persons (FDPs), the turmoil of this crisis is magnified significantly, and elevated pre-existing post-migration stressors and trauma-related mental health problems are acutely amplified. In a recent randomized control trial, Mindfulness-Based Trauma Recovery for Refugees (MBTR-R) led to large acute stress-buffering effects among Eritrean asylum seekers in Israel. The investigators thus developed Mindfulness-SOS for Refugees - a brief internet-based mobile-supported adaptation of the MBTR-R mental health intervention program - specifically designed to mitigate acute stress and related mental health symptoms among FDPs. The investigators will conduct a nonrandomized single-group intervention trial of the efficacy, safety, utilization, and related feasibility of Mindfulness-SOS for Refugees among a traumatized chronically stressed sample of East African asylum seekers in an urban post-displacement setting in the Middle East (Israel). The study will be carried out during an acutely stressful period of time for this population due to a COVID-19 pandemic national lockdown.

DETAILED DESCRIPTION:
Brief Background:

The COVID-19 pandemic is associated with a range of stressors and consequent mental health problems. For tens of millions of FDPs, stressors and sequelae of the pandemic are particularly magnified and severe, as their preexisting stress-related mental health problems are acutely exacerbated. In a recent randomized control trial prior to the COVID-19 pandemic, the investigators found significant therapeutic effects of MBTR-R - a 9-week, mindfulness- and compassion-based, trauma-sensitive, and socio-culturally adapted group intervention program designed for FDPs - for stress- and trauma-related mental health outcomes among Eritrean asylum seekers in Israel. In light of the COVID-19 pandemic, and to facilitate access, reach, and flexibility of mental health care among FDPs, the investigators developed Mindfulness-SOS for Refugees - a brief internet-based mobile-supported adaptation of the MBTR-R mental health intervention program - specifically designed to mitigate acute stress and related mental health symptoms among FDPs.

Study Aims:

Broadly, the study aims are: I) to test the efficacy of the Mindfulness-SOS for Refugees intervention program on stress- and trauma-related mental health outcomes (e.g. posttraumatic stress, depression), II) to test intervention safety - including rates of clinically significant deterioration in primary outcomes in response to the intervention, III) to assess participant utilization of the Mindfulness-SOS for Refugees intervention program, IV) to test whether Mindfulness-SOS for Refugees will lead to changes in targeted processes or mechanisms of change including mindful awareness and self-compassion, and V) to test whether expected pre-to-post intervention change in the targeted processes will predict expected pre-to-post intervention change in stress- and trauma-related mental health outcomes.

Study Overview:

Accordingly, the investigators will conduct a nonrandomized single-group intervention trial among a community sample of traumatized and chronically stressed East African asylum seekers (N=60, 50% female), residing in Israel in an urban post-displacement setting, during the COVID-19 pandemic. Over the course of three successive months, participants will be recruited from the community via public flyers, social networks, local non-governmental- (NGOs), and municipal- organizations working with FDPs. Participants will be assigned to Mindfulness-SOS for Refugees - a brief internet-based mobile-supported intervention program, entailing 8 brief sessions as well as 9 mindfulness meditation practice exercises - delivered via audio recordings using participants' personal smartphones. Over the course of the Mindfulness-SOS for Refugees intervention program, participants will receive administrative guidance (e.g. technical support in case of mobile phone and internet platform-related difficulties and relevant information of the internet-based mobile-supported intervention program and assessment); as well as adherence-focused guidance (e.g. adherence monitoring including weekly brief check-in telephone calls and smartphone text-based nudges to remind and prompt weekly adherence and assessment), in the participants' mother tongue, Tigrinya. Stress- and trauma-related mental health outcomes and targeted change processes will be assessed via self-report questionnaires pre-intervention, brief weekly assessments, and post-intervention. In addition to participants' self-report, participant-level utilization of the Mindfulness-SOS for Refugees intervention program will be digitally monitored. Participants will be encouraged to complete 2 sessions per week and practice each day for 4 weeks but can choose to extend this up to 8 weeks. Post-intervention assessments will be carried out when participants will complete the 8 sessions of the internet-based mobile-supported intervention program (recommended 4 weeks, a maximum of 8 weeks post-baseline, or when participants will indicate that they are no longer interested in participating in the intervention program). The intervention program and assessments will be completed on participants' smartphones.

ELIGIBILITY:
Inclusion Criteria:

* East African refugee or asylum seeker living in Israel
* Tigrinya fluency and literacy
* Owns a personal smartphone

Exclusion Criteria:

* Active suicidal ideation or/and past suicide attempt in the last year or/and passive suicidal ideation with clinical indicators of imminent suicide risk (e.g. severe paranoia)
* Current mental health treatment (i.e. psychotherapy or/and group therapy at least twice a month)
* Participation in the MBTR-R group in a previous study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Harvard Trauma Questionnaire according to DSM-5 (HTQ-5) | Change from immediately pre-intervention to 1-week post-intervention
  The Harvard Trauma Questionnaire according to DSM-5 (HTQ-5) is a 25-item self-report questionnaire to assess post-traumatic stress symptom severity (4-point Likert scale), with higher scores indicating greater levels of post-traumatic stress severity (minimum scale score 1 and maximum scale score 4), HTQ-5 mean cut-off score ≥ 2 is commonly used to identify categorical (diagnostic) symptom status of post-traumatic stress disorder
Brief Patient Health Questionnaire (PHQ-9) | Change from immediately pre-intervention to 1-week post-intervention
  The brief Patient Health Questionnaire (PHQ-9) is a 9-item self-report questionnaire to assess depression symptom severity (4-point Likert scale), with higher scores indicating greater levels of depression symptom severity (minimum scale score 0 and maximum scale score 27), PHQ-9 mean cut-off score ≥10 is commonly used to identify categorical (diagnostic) symptom status of depression
Beck's Anxiety Inventory (BAI) | Change from immediately pre-intervention to 1-week post-intervention
  6 Items of the Beck's Anxiety Inventory (BAI) self-report questionnaire will be used to assess anxiety symptom severity (4-point Likert scale), with higher scores indicating greater levels of anxiety symptom severity

SECONDARY OUTCOMES:
Post-Migration Living Difficulties Checklist (PMLD) | Change from immediately pre-intervention to 1-week post-intervention
  The Post-Migration-Living-Difficulties Checklist (PMLD) is a 9-item self-report questionnaire to assess post-migration stress (5-point Likert scale), with higher scores indicating greater levels of post-migration stress (minimum scale score 1 and maximum scale score 5)
Brief Inventory of Thriving (BIT) | Change from immediately pre-intervention to 1-week post-intervention
  One item of the Brief Inventory of Thriving (BIT) self-report questionnaire will be used to assess subjective well-being (5-point Likert scale), with higher scores indicating greater levels of subjective well-being
Dimensions of Anger Reactions-5 (DAR-5) | Change from immediately pre-intervention to 1-week post-intervention
  One item of the Dimensions of Anger Reactions-5 (DAR-5) self-report questionnaire will be used to assess anger duration (5-point Likert scale), with higher scores indicating greater levels of anger duration
Parenting Scale (PS) | Change from immediately pre-intervention to 1-week post-intervention
  One item of the Parenting Scale (PS) self-report questionnaire will be used to assess parental discipline strategies (5-point Likert scale), with higher scores indicating less effective discipline strategies
Modified 5-item Extended-Hurt/Insult/Threaten/Scream (Modified E-HITS) | Change from immediately pre-intervention to 1-week post-intervention
  One adapted item of the Modified 5-item Extended-Hurt/Insult/Threaten/Scream (Modified E-HITS) self-report questionnaire will be used to assess intimate partner violence (IPV) perpetration (5-point Likert scale), with higher scores indicating greater levels of perpetration of IPV
Positive and Negative Affect Schedule (PANAS) | Change from immediately pre-intervention to 1-week post-intervention, measured weekly up to 8 weeks
  The Positive and Negative Affect Schedule (PANAS) is a 20-item self-report questionnaire to assess positive and negative affect (5-point Likert scale), with higher scores indicating greater levels of activation of positively and negatively valanced affects
Brief assessment of mindful awareness | Change from immediately pre-intervention to 1-week post-intervention, measured weekly up to 8 weeks
  4 self-report Items will be used to assess mindful awareness (5-point Likert scale), with higher scores indicating greater levels of mindful awareness
Brief assessment of self-compassion | Change from immediately pre-intervention to 1-week post-intervention, measured weekly up to 8 weeks
  3 self-report Items will be used to assess self-compassion (5-point Likert scale), with higher scores indicating greater levels of self-compassion
Brief weekly assessment of formal and informal mindfulness practice | Weekly change from week 1 of intervention to 1-week post-intervention, up to 8 weeks
  2 self-report Items will be used to assess number of formal and informal mindfulness practice during the past week, with higher scores indicating greater number of mindfulness practices during the past week
Brief weekly assessment of post-traumatic stress | Weekly change from week 1 of intervention to 1-week post-intervention, up to 8 weeks
  4 self-report Items will be used to assess post-traumatic stress (5-point Likert scale), with higher scores indicating greater levels of post-traumatic stress
Brief weekly assessment of depression | Weekly change from week 1 of intervention to 1-week post-intervention, up to 8 weeks
  One self-report item will be used to assess depression (5-point Likert scale), with higher scores indicating greater levels of depression
Brief weekly assessment of anxiety | Weekly change from week 1 of intervention to 1-week post-intervention, up to 8 weeks
  One self-report item will be used to assess anxiety (5-point Likert scale), with higher scores indicating greater levels of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf, Tel Aviv, Central District, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zohar Puris S, Yuval K, Gebremariam G, Goldberg SB, Aviad N, Baldwin SA, Bernstein A. Nonrandomized Open Trial of a Mindfulness- and Compassion-Based Selective Preventive Mobile Health Intervention for Forcibly Displaced People. Mindfulness (N Y). 2025 Oct 2;16(10):2845-62. doi: 10.1007/s12671-025-02675-9. Online ahead of print. PMID 41050629
- [Derived] Blay Benzaken Y, Zohar S, Yuval K, Aizik-Reebs A, Gebremariam SG, Bernstein A. COVID-19 and Mental Health Among People Who Are Forcibly Displaced: The Role of Socioeconomic Insecurity. Psychiatr Serv. 2023 Feb 1;74(2):158-165. doi: 10.1176/appi.ps.202200052. Epub 2022 Jul 14. PMID 35833254
- See also: Mindfulness-SOS for Refugees intervention program study website — https://www.mindfulness-sos-study.com/